CLINICAL TRIAL: NCT04766554
Title: A Multicenter, Randomized, Controlled Clinical Trial of Cerebral Oxygen Saturation Monitoring In Cardiac Surgery (COSMICS)
Brief Title: Cerebral Oxygen Saturation Monitoring In Cardiac Surgery (COSMICS)
Acronym: COSMICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia de Laranjeiras (Other)
Responsible Party: Principal Investigator, Carlos Galhardo Jr., Chief of Adult Cardiac Anesthesia Division, Instituto Nacional de Cardiologia de Laranjeiras
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COSMICS STUDY
Record Dates: First submitted 2021-02-16; First posted 2021-02-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Disease; Cognitive Dysfunction
Keywords: Intraoperative Neurophysiologic Monitorings
MeSH Terms: conditions — Heart Diseases; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Patients will be monitored with cerebral oximetry using INVOS 5100 monitor (Covidien, Boulder, CO), with electrodes applied bilaterally in the frontal region. Following the placement of the electrodes, the baseline records HR, blood pressure, rSO2, and peripheral O2 saturation (SPO2) will be recorded following 1 minute of electrode placement and the proper verification of the signal on the monitor. Later, during the surgery, if the rSO2 reaches levels below 15% of the baseline values or below 50% in absolute value for over 30 seconds, protocol-based interventions will be performed in the intervention group to return the oximeter to baseline values. The alarm on the equipment should be programmed to signal values below 15% of the baseline values.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be masked concerning the allocation group. The anesthesiologist responsible for conducting the case will not be involved in the application of the neurocognitive tests, nor will he be aware of the test results. Investigators who apply the tests will be covered up by the patient allocation group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebral Oxymetry Monitoring (Active Comparator): The following procedures should be performed sequentially in the event of cerebral desaturation after 30 seconds:
  1. The positioning of the head, the presence of facial plethora, and bad position of catheters should be corrected;
  2. In case of arterial hypotension, the causal factors should be assessed and treated;
  3. In the presence of arterial hypoxemia, the causal factors should be assessed and treated to maintain a PaO2 > 150 mmHg;
  4. In the presence of hypercapnia, adjust the ventilation parameters avoiding hyperventilation;
  5. In the presence of anemia, the causal factors should be assessed, and the decision to undergo transfusion should also take into consideration the presence of tissue hypoperfusion;
  6. In cases of SvO2 below 70% and signs of hemodynamic instability, optimize fluid replacement and ventricular global contractility;
  7. Assess the increase of brain consumption of O2, avoiding the superficial level of anesthesia, hyperthermia, and tremors.
  Interventions: Device: Cerebral oximetry monitor (The INVOS® Cerebral/Somatic Oximeter) and protocol-based interventions
- Control Group (No Intervention): Patients will be treated according to the attending anesthesiologist, without the monitoring of cerebral oximetry, but to maintain a heart rate between 70 - 100 bpm, lactate levels <3 mmol/L and urine output> 0.5mL/Kg/h. In case of arterial hypotension the causal factors should be assessed and treated; in case of SvO2 below 70% and signs of hemodynamic instability, optimize volume replacement and global ventricular contractility through inotropic agents (epinephrine, dobutamine or milrinone); in the presence of anemia (Hb <6 to 7g/dL during CPB or Hb <8g/dL in the pre-CPB or post-CPB period), the causal factors should be assessed and the decision to transfuse should also take into account the presence of hypoperfusion tissue (increased lactate, low SvO2, acidosis); in episodes of bradycardia with hemodynamic instability, atropine may be used.

INTERVENTIONS:
Device: Cerebral oximetry monitor (The INVOS® Cerebral/Somatic Oximeter) and protocol-based interventions — In the intervention group, an alarm threshold below 15% of the baseline rSO2 value will be established. Based on the predetermined algorithm the rSO2 will be maintained at or above 85% of the baseline measurements. If the rSO2 reaches levels below 15% of the baseline values or below 50% in absolute value for over 30 seconds, protocol-based interventions will be performed to restore rSO2 to baseline levels.
  Arms: Cerebral Oxymetry Monitoring

SUMMARY:
Neurological dysfunction continues to be one of the complications of considerable concern in patients undergoing cardiac surgery. It was previously reported in the literature, that cerebral oxygen desaturation during cardiac surgery was associated with an increased incidence of cognitive impairment. This study aims to determine whether continuous monitoring of cerebral oximetry improves the neurocognitive outcome in coronary artery bypass surgery when associated with predetermined intervention protocol to optimize cerebral oxygenation.

DETAILED DESCRIPTION:
Despite all the progress over the last decades regarding the improvement of the perioperative care of patients with heart disease and the development of new surgical techniques, neurological dysfunction continues to be one of the complications of the greatest concern in patients undergoing cardiac surgery with cardiopulmonary bypass. Brain injury can manifest itself through permanent or temporary injury, contributing to the increase in-hospital mortality, in the length of stay in intensive care, in the length of hospital stay, to a higher incidence of motor dysfunction requiring rehabilitation, and consequently, to reduced quality of life.

Even though the causes of brain injury are multifactorial, perioperative cerebral hypoperfusion, tissue hypoxia, and thromboembolic events are among the main factors related to neurological dysfunction.

Several clinical studies have indicated an association between cerebral desaturation and the increase of neurological complications. Cerebral oximetry monitoring using near-infrared spectroscopy (NIRS) is a non-invasive technique used to estimate regional cerebral oxygen saturation (rSO2) and has been associated with diminishing the incidence of neurological complications.

There is no consensus in the literature about its real benefit, mainly due to the absence of well-designed scientific studies that demonstrate that cerebral desaturation associated with intervention measures to improve rSO2, are related to the prevention of neurological dysfunction in adult cardiac surgery.

The study hypothesis evaluates whether continuous monitoring of cerebral oximetry improves the neurocognitive outcome in coronary artery bypass surgery when associated with early interventions to optimize rSO2.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older
* Elective coronary artery bypass graft surgery using cardiopulmonary bypass
* Preoperative cognitive assessment by means of Mini-Mental State Examination (MMSE) test, greater than or equal to 24
* Signed informed consent

Exclusion Criteria:

* Patients with focal neurologic deficit
* Carotid artery stenosis greater than 70%
* Patients with pre-existing cognitive dysfunction
* Patients with psychotic disorders
* History of allergy to adhesive part of the electrode
* History of craniofacial surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Preoperative cognitive function | Pre-surgery (within 10 days before)
  Mini Mental State Examination (MMSE)
Postoperative cognitive dysfunction - delayed cognitive recovery | Post-surgery (7 days after surgery)
  Mini Mental State Examination (MMSE)
Postoperative cognitive dysfunction - neurocognitive disorder | Post-surgery (90 days after surgery)
  Mini Mental State Examination (MMSE)
Preoperative cognitive function II | Pre-surgery (within 10 days before)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - delayed cognitive recovery II | Post-surgery (7 days after surgery)
  Montreal Cognitive Assessment (MoCA) test
Postoperative cognitive dysfunction - neurocognitive disorder II | Post-surgery (90 days after surgery)
  Montreal Cognitive Assessment (MoCA) test
Preoperative cognitive function III | Pre-surgery (within 10 days before)
  The Telephone Interview for Cognitive Status (TICS)
Postoperative cognitive dysfunction - delayed cognitive recovery III | Post-surgery (7 days after surgery)
  The Telephone Interview for Cognitive Status (TICS)
Postoperative cognitive dysfunction - neurocognitive disorder III | Post-surgery (90 days after surgery)
  The Telephone Interview for Cognitive Status (TICS)

SECONDARY OUTCOMES:
Incidence of postoperative delirium | Delirium assessment CAM-ICU preoperatively (baseline) and postoperatively twice a day during the first seven days or until discharge
  Delirium will be assessed postoperatively for seven days or until discharge
Neurological injury type I (stroke) | Post-surgery (until 30 days after surgery)
  The incidence of neurological injury type I will be evaluated for 30 days
Duration of mechanical ventilation | Post-surgery (until 30 days after surgery)
  The duration of mechanical ventilation will be evaluated
Length of stay at the intensive care unit (ICU) | Post-surgery (until 30 days after surgery)
  The length of stay at the intensive care unit (ICU) will be evaluated
Length of stay at the hospital | Post-surgery (until 30 days after surgery)
  The length of stay at the hospital will be evaluated
Incidence of mortality resulting from all causes | Post-surgery (until 30 days after surgery)
  All causes of mortality will be assessed for 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Galhardo, MD, Principal Investigator — Instituto Nacional de Cardiologia
Locations (2):
- Brazil (2):
  - Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro
  - Hospital São José, Criciúma, Santa Catarina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zheng F, Sheinberg R, Yee MS, Ono M, Zheng Y, Hogue CW. Cerebral near-infrared spectroscopy monitoring and neurologic outcomes in adult cardiac surgery patients: a systematic review. Anesth Analg. 2013 Mar;116(3):663-76. doi: 10.1213/ANE.0b013e318277a255. Epub 2012 Dec 24. PMID 23267000
- [Result] Deschamps A, Hall R, Grocott H, Mazer CD, Choi PT, Turgeon AF, de Medicis E, Bussieres JS, Hudson C, Syed S, Seal D, Herd S, Lambert J, Denault A, Deschamps A, Mutch A, Turgeon A, Denault A, Todd A, Jerath A, Fayad A, Finnegan B, Kent B, Kennedy B, Cuthbertson BH, Kavanagh B, Warriner B, MacAdams C, Lehmann C, Fudorow C, Hudson C, McCartney C, McIsaac D, Dubois D, Campbell D, Mazer D, Neilpovitz D, Rosen D, Cheng D, Drapeau D, Dillane D, Tran D, Mckeen D, Wijeysundera D, Jacobsohn E, Couture E, de Medicis E, Alam F, Abdallah F, Ralley FE, Chung F, Lellouche F, Dobson G, Germain G, Djaiani G, Gilron I, Hare G, Bryson G, Clarke H, McDonald H, Roman-Smith H, Grocott H, Yang H, Douketis J, Paul J, Beaubien J, Bussieres J, Pridham J, Armstrong JN, Parlow J, Murkin J, Gamble J, Duttchen K, Karkouti K, Turner K, Baghirzada L, Szabo L, Lalu M, Wasowicz M, Bautista M, Jacka M, Murphy M, Schmidt M, Verret M, Perrault MA, Beaudet N, Buckley N, Choi P, MacDougall P, Jones P, Drolet P, Beaulieu P, Taneja R, Martin R, Hall R, George R, Chun R, McMullen S, Beattie S, Sampson S, Choi S, Kowalski S, McCluskey S, Syed S, Boet S, Ramsay T, Saha T, Mutter T, Chowdhury T, Uppal V, Mckay W; Canadian Perioperative Anesthesia Clinical Trials Group. Cerebral Oximetry Monitoring to Maintain Normal Cerebral Oxygen Saturation during High-risk Cardiac Surgery: A Randomized Controlled Feasibility Trial. Anesthesiology. 2016 Apr;124(4):826-36. doi: 10.1097/ALN.0000000000001029. PMID 26808629
- [Result] Slater JP, Guarino T, Stack J, Vinod K, Bustami RT, Brown JM 3rd, Rodriguez AL, Magovern CJ, Zaubler T, Freundlich K, Parr GV. Cerebral oxygen desaturation predicts cognitive decline and longer hospital stay after cardiac surgery. Ann Thorac Surg. 2009 Jan;87(1):36-44; discussion 44-5. doi: 10.1016/j.athoracsur.2008.08.070. PMID 19101265
- [Result] Lei L, Katznelson R, Fedorko L, Carroll J, Poonawala H, Machina M, Styra R, Rao V, Djaiani G. Cerebral oximetry and postoperative delirium after cardiac surgery: a randomised, controlled trial. Anaesthesia. 2017 Dec;72(12):1456-1466. doi: 10.1111/anae.14056. Epub 2017 Sep 22. PMID 28940368
- [Result] Colak Z, Borojevic M, Bogovic A, Ivancan V, Biocina B, Majeric-Kogler V. Influence of intraoperative cerebral oximetry monitoring on neurocognitive function after coronary artery bypass surgery: a randomized, prospective study. Eur J Cardiothorac Surg. 2015 Mar;47(3):447-54. doi: 10.1093/ejcts/ezu193. Epub 2014 May 7. PMID 24810757
- [Result] Serraino GF, Murphy GJ. Effects of cerebral near-infrared spectroscopy on the outcome of patients undergoing cardiac surgery: a systematic review of randomised trials. BMJ Open. 2017 Sep 7;7(9):e016613. doi: 10.1136/bmjopen-2017-016613. PMID 28882917
- [Result] Murkin JM, Adams SJ, Novick RJ, Quantz M, Bainbridge D, Iglesias I, Cleland A, Schaefer B, Irwin B, Fox S. Monitoring brain oxygen saturation during coronary bypass surgery: a randomized, prospective study. Anesth Analg. 2007 Jan;104(1):51-8. doi: 10.1213/01.ane.0000246814.29362.f4. PMID 17179242